CLINICAL TRIAL: NCT00927004
Title: A Randomised Placebo-controlled Trail of Mechanical and Cold Hyperalgesia in Subjects With Painful Knee Osteoarthritis, Compared With Matched Controls, & Whether This Hyperalgesia Can be Modified by a 2-week Course of Etoricoxib 60mg.
Brief Title: Efficacy of Etoricoxib 60 mg in Modifying Pain Hypersensitivity in People With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Curtin University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Penny Moss, Lecturer, Curtin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Moss IISP#36409; 3144 Wright-Merck; HR47-2009
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis; Pain
Keywords: mechanical hyperalgesia; cold hyperalgesia; chronic pain
MeSH Terms: conditions — Osteoarthritis; Pain; Hyperalgesia; Chronic Pain | interventions — Etoricoxib; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib 60 mg (Experimental)
  Interventions: Drug: Etoricoxib (Arcoxia)
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Etoricoxib (Arcoxia) — 60 mg, daily dose, oral delivery, 14 days duration
  Other Names: Arcoxia
  Arms: Etoricoxib 60 mg
Drug: Sugar pill — Daily dose (1 pill), oral delivery, 14 days
  Arms: Sugar pill

SUMMARY:
This study aims to better understand the way in which painful osteoarthritis affects different people and whether an anti-inflammatory medication such as Arcoxia (etoricoxib) can help to modify this pain. The study will use questionnaires and tests of pain sensitivity to identify arthritis sufferers with more widespread, nerve-type pain and then to investigate whether a daily dose of Arcoxia is more effective than a placebo pill in reducing these symptoms and improving functional movements. The study will also be comparing the same test results of a small group of subjects without knee pain.

ELIGIBILITY:
Inclusion Criteria:

* unilateral diagnosis of Knee OA > 6 months
* knee pain > 4/10 on WOMAC pain subscale
* if pain in contralateral knee, no greater than "mild"
* no other significant joint involvement
* ARA functional Class I, II or III
* no arthroscopy or injections into index knee in last 6 months

Exclusion Criteria:

* history of systemic inflammatory or chronic pain disorders (especially fibromyalgia)
* neurological deficit
* recent (< 6 months) lower limb surgery
* allergic reaction to NSAIDs or aspirin
* skin allergies, dermatitis
* contraindications to Cox-2 inhibitors:

  * congestive heart failure (NYHA II-IV)
  * unstable hypertension
  * ischaemic heart disease
  * peripheral artery disease
  * cerebrovascular disease including CABG or angioplasty within 1 year
* severe hepatic dysfunction
* active GI bleeding or peptic ulceration
* reduced creatinine clearance < 30 mL/min
* current use of high dose (> 325 mg daily) aspirin

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | 15 days, 3 days
Western Ontario and McMaster University Osteoarthritis Index (knee) - pain subscale | 15 days, 3 days

SECONDARY OUTCOMES:
Cold Pain Threshold | 15 days, 3 days
Topical Cold Response | 15 days, 3 days
Functional Measure (aggregated locomotor score, sit-to-stand time) | 15 days, 3 days
WOMAC (knee) total | 15 days, 3 days
SF-36v2 | 15 days, 3 days
Pain Quality Assessment Scale | 15 days, 3 days
PainDETECT questionnaire | 15 days, 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Tony Wright, PhD, Principal Investigator — Curtin University
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Moss P, Benson HAE, Will R, Wright A. Fourteen days of etoricoxib 60 mg improves pain, hyperalgesia and physical function in individuals with knee osteoarthritis: a randomized controlled trial. Osteoarthritis Cartilage. 2017 Nov;25(11):1781-1791. doi: 10.1016/j.joca.2017.07.009. Epub 2017 Aug 2. PMID 28778815